CLINICAL TRIAL: NCT03650231
Title: Comparison of Abbott Architect®, Siemens Immulite®, and Diasorin Liaison® for Determination of Epstein-Barr Virus Serological Diagnosis
Brief Title: Comparison of Technics for Determination of Epstein-Barr Virus Serological Diagnosis
Acronym: DIAGEPS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0042
Record Dates: First submitted 2018-08-22; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: EBV
Keywords: Epstein-barr virus; infectious mononucleosis
MeSH Terms: conditions — Epstein-Barr Virus Infections; Infectious Mononucleosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Serological giagnosis — The serological diagnosis of EBV infection was performed in the Amiens University Hospital virology laboratory (France). 91 routinely collected samples were analyzed by Immulite, Architect, and Liaison Blood samples were centrifuged for 15 min at 2500g at room temperature. Sera were aliquoted and first analyzed by Immulite. All samples were tested for EBV VCA IgG, EBV VCA IgM and EBV EBNA IgG in order to determine infection status (primary EBV infection, past infection, absence of infection and indeterminate status).

SUMMARY:
This study compared the performance of three automated immunoassays, Architect (Abbott), Immulite (Siemens) and Liaison (Diasorin), for Epstein-Barr virus (EBV) serology. Ninety-one serum samples collected in Amiens University Hospital were analyzed for the presence of Viral Capsid Antigen (VCA) IgG and IgM and Epstein-Barr Nuclear Antigen (EBNA) IgG. The agreement between the three assays was calculated for each marker individually and for determination of the EBV profile, based on interpretation of the combination of these three EBV markers.

DETAILED DESCRIPTION:
This retrospective study was conducted on 91 samples collected between 2014 and 2015 for which EBV diagnosis was requested. The serological diagnosis of EBV infection was performed in the Amiens University Hospital virology laboratory (France). The median age of patients was 34 years (mean: 38 years, range: 3-82 year) with a sex ratio of 50%. Sixteen of the 91 samples concerned children (<15 years).

This study compared the performance of three automated immunoassays, Architect (Abbott), Immulite (Siemens) and Liaison (Diasorin), for Epstein-Barr virus (EBV) serology. Ninety-one serum samples collected in Amiens University Hospital were analyzed for the presence of Viral Capsid Antigen (VCA) IgG and IgM and Epstein-Barr Nuclear Antigen (EBNA) IgG. The agreement between the three assays was calculated for each marker individually and for determination of the EBV profile, based on interpretation of the combination of these three EBV markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with EBV diagnosis
* Age between 3 and 82 years

Exclusion Criteria:

* Patient <3 years
* Patient > 82 years

Ages: 3 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 91 samples collected between 2014 and 2015 for which EBV diagnosis was requested. The serological diagnosis of EBV infection was performed in the Amiens University Hospital virology laboratory (France). The median age of patients was 34 years (mean: 38 years, range: 3-82 year) with a sex ratio of 50%. Sixteen of the 91 samples concerned children (<15 years)
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-10-29 (Actual); Study Completion 2017-10-29 (Actual)

PRIMARY OUTCOMES:
Capacity of the three assays to detect VCA IgM | 2years
  The aim of the present study is to evlaute the capacity of the three tests to detect VCA IgM. 91 samples was collected and tested for EBV VCA IgG, EBV VCA IgM and EBV EBNA IgG in order to determine infection status (primary EBV infection, past infection, absence of infection and indeterminate status).

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Castelain, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No